CLINICAL TRIAL: NCT06037798
Title: The Cranio-cervical Flexion Test, Using the NOD. A Pilot and Feasibility Study
Brief Title: The Cranio-cervical Flexion Test Using the NOD Device
Acronym: CCFT-NOD
Status: Completed | Type: Observational
Sponsor: Zurich University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Markus J. Ernst, Principal investigator, Zurich University of Applied Sciences
Other Study IDs: CCFT-NOD
Record Dates: First submitted 2023-08-30; First posted 2023-09-14 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Muscle Strength; Neck Muscle Issue; Bruxism; EMG
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bruxism: subjects with known bruxism, no TMD, primary headache or neck pain
  Interventions: Other: cranio-cervical flexion test with NOD
- healthy: non-bruxism, no primary headache, TMD or neck pain
  Interventions: Other: cranio-cervical flexion test with NOD

INTERVENTIONS:
Other: cranio-cervical flexion test with NOD — testing the anterior neck muscles during a nodding movement and by using a dynamometer

SUMMARY:
to measure strength of the deep anterior neck muscles with a new measurement protocol and by using the NOD device, a dynamometer, in subjects with and without bruxism, and compared to EMG on the superficial muscles of the anterior neck and the masseter muscle.

ELIGIBILITY:
Inclusion Criteria:

* with or without bruxism
* German fluent
* informend consent

Exclusion Criteria:

* primary headache
* cranio-mandibulary disorders (CMD) in >3 months within the last 12 months
* current neck pain intensity > 2 out of 10 on Numeric rating scale
* known:
* neurological pathologies
* mental impairments or diseases
* pregnancy
* rheumatic disorders

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult subjects with and without bruxism
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
activation score = AS | baseline
  stepwise (5 steps) and correct (no substitution by the superficial muscles) activation of the deep neck flexors, that can be hold for 10 seconds: Each step increases by 3.4N. The scale will be offset, starting at 0N. Steps are accordingly: 3.4N, 6.8N, 10.2N, 13.6N, 17N. Higher scores denote better function
performance index= PI | baseline
  number of correctly performed 10 second holds at each incremental step. number between 1 and 10. Higher scores denote better function.

SECONDARY OUTCOMES:
Neck-Pain | baseline
  neck pain, headache or discomfort during or immediate after the test protocol, measured by a numeric rating scale from 0 to 10. Higher scores denote more pain or discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- Zurich University of applied sciences, Winterthur, Switzerland

IPD SHARING:
Plan to Share IPD: No
data can be shared on demand

REFERENCES:
- [Background] Ernst MJ, Sax N, Meichtry A, Aegerter AM, Luomajoki H, Ludtke K, Gallina A, Falla D; NEXpro collaboration group. Cervical musculoskeletal impairments and pressure pain sensitivity in office workers with headache. Musculoskelet Sci Pract. 2023 Aug;66:102816. doi: 10.1016/j.msksp.2023.102816. Epub 2023 Jun 26. PMID 37394322
- [Background] Chiu TT, Law EY, Chiu TH. Performance of the craniocervical flexion test in subjects with and without chronic neck pain. J Orthop Sports Phys Ther. 2005 Sep;35(9):567-71. doi: 10.2519/jospt.2005.35.9.567. PMID 16268243
- [Background] James G, Doe T. The craniocervical flexion test: intra-tester reliability in asymptomatic subjects. Physiother Res Int. 2010 Sep;15(3):144-9. doi: 10.1002/pri.456. PMID 20146239
- [Background] Jull G, Amiri M, Bullock-Saxton J, Darnell R, Lander C. Cervical musculoskeletal impairment in frequent intermittent headache. Part 1: Subjects with single headaches. Cephalalgia. 2007 Jul;27(7):793-802. doi: 10.1111/j.1468-2982.2007.01345.x. PMID 17598761
- [Result] Carrasco-Uribarren A, Marimon X, Portela A, Cabanillas-Barea S, Rodriguez-Rubio PR, Perez RA. A Novel Device for Assessment and Treatment of Upper Cervical Spine: Test-Retest Reliability Study. J Clin Med. 2023 Mar 1;12(5):1954. doi: 10.3390/jcm12051954. PMID 36902739
- [Result] Romeo A, Baccini M, Carreras G, Sagripanti M, Ruggeri M, Pillastrini P, Di Bari M. Reliability, Validity, and Responsiveness of the Craniocervical Flexion Test in People Who Are Asymptomatic and Patients With Nonspecific Neck Pain: A Systematic Review and Meta-Analysis. Phys Ther. 2022 Jul 4;102(7):pzac054. doi: 10.1093/ptj/pzac054. PMID 35554598
- [Result] Selistre LFA, Melo CS, Noronha MA. Reliability and Validity of Clinical Tests for Measuring Strength or Endurance of Cervical Muscles: A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2021 Jun;102(6):1210-1227. doi: 10.1016/j.apmr.2020.11.018. Epub 2020 Dec 28. PMID 33383030